CLINICAL TRIAL: NCT02324374
Title: The Role of in Vivo Real Time Endocytoscopy in Diagnosing Colorectal Neoplasia
Brief Title: Endocytoscopy and Colorectal Neoplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 813061
Record Dates: First submitted 2014-12-18; First posted 2014-12-24 (Estimated); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Colon Cancer
Keywords: colon cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (1):
- Endocytoscopy During Colonoscopy (Experimental): Colonoscopies will be performed as per routine practice. When a colorectal lesion is found that would normally require biopsy or polypectomy; the lesion will be evaluated by chromoendoscopy with the application of 10 ml 1% methylene blue followed by the inspection with the endocytoscope at both magnifications (450X and 1100X). The endocytoscopic images of the abnormal area will be recorded prior to biopsy or removal of the suspicious tissue. For each lesion, a matching endocytoscopy image from normal adjacent tissue will also be obtained, at least 5cm away from the suspect site, but within the same segment of intestine (e.g. ascending colon). No biopsy will be obtained from normal tissue, and this will be assumed to be normal. Following image acquisition, the lesion will be biopsied or removed as per standard clinical care.
  Interventions: Device: Endocystoscopy During Colonoscopy; Device: Endocytoscope

INTERVENTIONS:
Device: Endocystoscopy During Colonoscopy — Colonoscopies will be performed as per routine practice. When a colorectal lesion is found that would normally require biopsy or polypectomy; the lesion will be evaluated by chromoendoscopy with the application of 10 ml 1% methylene blue followed by the inspection with the endocytoscope at both magnifications (450X and 1100X). The endocytoscopic images of the abnormal area will be recorded prior to biopsy or removal of the suspicious tissue. For each lesion, a matching endocytoscopy image from normal adjacent tissue will also be obtained, at least 5cm away from the suspect site, but within the same segment of intestine (e.g. ascending colon). No biopsy will be obtained from normal tissue, and this will be assumed to be normal. Following image acquisition, the lesion will be biopsied or removed as per standard clinical care.
  Other Names: endocytoscope
Device: Endocytoscope — The endocytoscopes, prototype I and prototype II will be used during the study along with the standard colonoscopes. The endocytoscope is a soft catheter type endoscope, with an outside diameter of 3.4 mm at the distal end and 3.2 at the shaft, and total length of 380 cm (working length of 250 cm) which uses a lens system for magnification. The Prototype 1 endocytoscope (low resolution type) has a magnification capability of x 450, depth of field of 50 um, field of view of 300X 300 um with a spatial resolution of 1.7 um. The Prototype 2 (high resolution) has a magnification capability of x1125, depth of field of 5um, field of view of 120X 120 um, and a spatial resolution of 4.2 um, The ECS system can be passed through the working channel of a standard colonoscope.

SUMMARY:
This will be a feasibility study to evaluate the role of endocytoscopy in classifying colorectal polyps in vivo. The primary outcomes will be to determine the key endocytoscopy image features of neoplastic and non-neoplastic colorectal polyps. The target population will include adult subjects undergoing screening and surveillance colonoscopies.

DETAILED DESCRIPTION:
Colorectal cancer has been recognized as the second most common cause of cancer related death in the US (1). Most colorectal cancers arise from adenomatous polyps that progress. Colon polyps are usually classified as neoplastic (adenoma and carcinoma) and non-neoplastic (most commonly hyperplastic). Standard endoscopic inspection cannot reliably distinguish between polyp types. Thus, all visualized polyps during standard colonoscopies are typically removed. Since almost half of all polyps are hyperplastic, a large proportion of unnecessary polypectomies increase the time, risk, and cost of colonoscopies.

Various studies have showed improved diagnostic accuracy of different types of polyps when broad field techniques such as chromoendoscopy with the use of topical stains were used to detect and characterize lesions (2-4). Chromoendoscopy, though an approved method of lesion characterization during endoscopic evaluation of colorectal lesions, is time consuming and non-standardized. Recently small field techniques such as confocal microscopy and endocytoscopy have been introduced enabling visualization of the gastrointestinal tract at a cellular level, thus allowing diagnosis and classification of colorectal lesions in vivo.

Confocal endomicroscopy used along with chromoendoscopy to detect and characterize lesions has been studied extensively and reported to have a high accuracy in diagnosing neoplastic and nonneoplastic lesions of the gastrointestinal tract (5-12). One of the major limitations of the confocal system is the mandatory use of dyes such as topical Acriflavine or intravenous Fluorescein. However, there are issues with the application of these dyes; the risk of DNA damage with Acriflavine reduced its use. In addition, although intravenous fluorescein is FDA approved for diagnostic fluorescein angiography, its gastrointestinal application is an off-label indication and considered class IIb by the FDA. The other major limitation of the current confocal system is that it requires a dedicated confocal endoscope marketed by a single manufacturer. Thus, the use of confocal imaging requires purchase of specific confocal endoscopes.

Endocytoscopy is based on the technology of light-contact microscopy. The current endocytoscopy system (ECS) consists of two prototypes; Prototype one gives a low magnification (XEC300) with a maximal 450X magnification and field of view of 300X300 um, Prototype two provide a high magnification (XEC120) with a maximal 1100X magnification and a field of view of 120X120 um. In contrast to confocal endomicroscopy, the endocytoscopes can be easily passed through an accessory channel of the conventional therapeutic endoscope. This method does not require the use of intravenous contrast agents. Instead, it uses topical staining such as methylene blue or crestyl violet, which is applied routinely to facilitate visualization and removal of advanced colorectal polyps through endoscopic mucosal resection during colonoscopy.

The endocytoscopy system has only recently been introduced and hence there are very few studies reporting its use.

A prospective study from Japan used endocytoscopy on 113 patients to obtain real time histological images in vivo during colonoscopy (13). With the ECS system, it was possible to observe lesions at the cellular level, evaluate cellular atypia and distinguish between neoplastic and nonneoplastic lesions when compared to histology which was used as the gold standard. The correlation between the endocytoscopic and histological diagnosis was statistically significant. Eleber et al (14) also reported a sensitivity and specificity of 79% and 90 %, respectively of the ECS system in diagnosing neoplastic lesions in 28 patients with colonic lesions. Furthermore the study by Cipoletta et al (15) demonstrated that the ECS system provides real time imaging in vivo with clear visualization of cellular details and features of dysplasia of aberrant crypt foci, considered to be the earliest precursor of colorectal cancer. In addition Rotondano et al (15) also confirmed high positive predictive values for diagnosing hyperplastic polyps as well as dysplastic polyps including low, high grade dysplasia as well as invasive cancer.

A recent systematic review of all published studies also confirmed that endocytoscopy is a safe and effective new endoscopic imaging technique to obtain in vivo histology and guided biopsies with high diagnostic accuracy (17).

No associated risks related to the endocystoscopy procedures have been reported in all published studies (12-17).

This specific diagnostic tool of in vivo histology with the use of high resolution endocytoscopy system would allow endoscopists to perform targeted biopsies and in some cases (if warranted based on the in vivo images) to proceed directly to endoscopic resection of lesions. It may also guide assessment of the completeness of the endoscopic intervention with detection of any residual neoplastic tissue at the index exam as well as on follow up colonoscopy exams. Other potential benefits include elimination of random biopsies for surveillance of mucosal disease, elimination of sampling error, limitation of unnecessary polypectomies, hence ultimately resulting in cost effectiveness and improved patient outcomes.

In summary, endocytoscopy has the potential to fundamentally change the way endoscopy and pathology interact by allowing near histological quality imaging in vivo, without the need, risk, and cost of tissue removal.

ELIGIBILITY:
Inclusion Criteria:

• Age above 18, any patient undergoing screening or surveillance colonoscopy.

Exclusion Criteria:

* Pregnancy
* Unwillingness to consent
* Lack of any pathological state that would require biopsy at the time of endoscopy (will be considered "screen failure" since this will not be known until after consent is obtained and sedated endoscopy performed).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-06; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Unblinded Analysis of Endocytoscopic Images of Colorectal Lesions (Technical quality of the images will be compared to histology and rated on a scale of 1-5 (1-worst, 3- acceptable, 5-being equal to histology) | 30 Days (from Colonoscopy)
  Endocytoscopic images of colorectal lesions will be reviewed in an unblinded fashion, in a group of 10 side by side images, by the endoscopists (AMB, NA) and the pathologist (AS). Technical quality of the images will be compared to histology and rated on a scale of 1-5 (1-worst, 3- acceptable, 5-being equal to histology). Only images with a score of 3 or better will be used for analysis. The percentage of cases with at least one adequate image per site will be described. The basic characteristics of images allowing distinction between neoplastic, non-neoplastic and normal tissue will be established.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Hawk ET, Levin B. Colorectal cancer prevention. J Clin Oncol. 2005 Jan 10;23(2):378-91. doi: 10.1200/JCO.2005.08.097. PMID 15637400
- [Background] Hurlstone DP, Fujii T, Lobo AJ. Early detection of colorectal cancer using high-magnification chromoscopic colonoscopy. Br J Surg. 2002 Mar;89(3):272-82. doi: 10.1046/j.0007-1323.2001.02040.x. PMID 11872049
- [Background] Hurlstone DP, Cross SS, Slater R, Sanders DS, Brown S. Detecting diminutive colorectal lesions at colonoscopy: a randomised controlled trial of pan-colonic versus targeted chromoscopy. Gut. 2004 Mar;53(3):376-80. doi: 10.1136/gut.2003.029868. PMID 14960519
- [Background] Kiesslich R, Fritsch J, Holtmann M, Koehler HH, Stolte M, Kanzler S, Nafe B, Jung M, Galle PR, Neurath MF. Methylene blue-aided chromoendoscopy for the detection of intraepithelial neoplasia and colon cancer in ulcerative colitis. Gastroenterology. 2003 Apr;124(4):880-8. doi: 10.1053/gast.2003.50146. PMID 12671882
- [Background] Kiesslich R, Burg J, Vieth M, Gnaendiger J, Enders M, Delaney P, Polglase A, McLaren W, Janell D, Thomas S, Nafe B, Galle PR, Neurath MF. Confocal laser endoscopy for diagnosing intraepithelial neoplasias and colorectal cancer in vivo. Gastroenterology. 2004 Sep;127(3):706-13. doi: 10.1053/j.gastro.2004.06.050. PMID 15362025
- [Background] Sakashita M, Inoue H, Kashida H, Tanaka J, Cho JY, Satodate H, Hidaka E, Yoshida T, Fukami N, Tamegai Y, Shiokawa A, Kudo S. Virtual histology of colorectal lesions using laser-scanning confocal microscopy. Endoscopy. 2003 Dec;35(12):1033-8. doi: 10.1055/s-2003-44595. PMID 14648417
- [Background] Polglase AL, McLaren WJ, Skinner SA, Kiesslich R, Neurath MF, Delaney PM. A fluorescence confocal endomicroscope for in vivo microscopy of the upper- and the lower-GI tract. Gastrointest Endosc. 2005 Nov;62(5):686-95. doi: 10.1016/j.gie.2005.05.021. PMID 16246680
- [Background] Kiesslich R, Goetz M, Lammersdorf K, Schneider C, Burg J, Stolte M, Vieth M, Nafe B, Galle PR, Neurath MF. Chromoscopy-guided endomicroscopy increases the diagnostic yield of intraepithelial neoplasia in ulcerative colitis. Gastroenterology. 2007 Mar;132(3):874-82. doi: 10.1053/j.gastro.2007.01.048. Epub 2007 Jan 31. PMID 17383417
- [Background] Kiesslich R, Gossner L, Goetz M, Dahlmann A, Vieth M, Stolte M, Hoffman A, Jung M, Nafe B, Galle PR, Neurath MF. In vivo histology of Barrett's esophagus and associated neoplasia by confocal laser endomicroscopy. Clin Gastroenterol Hepatol. 2006 Aug;4(8):979-87. doi: 10.1016/j.cgh.2006.05.010. Epub 2006 Jul 13. PMID 16843068
- [Background] Kiesslich R, Hoffman A, Goetz M, Biesterfeld S, Vieth M, Galle PR, Neurath MF. In vivo diagnosis of collagenous colitis by confocal endomicroscopy. Gut. 2006 Apr;55(4):591-2. doi: 10.1136/gut.2005.084970. No abstract available. PMID 16531549
- [Background] Kiesslich R, Goetz M, Burg J, Stolte M, Siegel E, Maeurer MJ, Thomas S, Strand D, Galle PR, Neurath MF. Diagnosing Helicobacter pylori in vivo by confocal laser endoscopy. Gastroenterology. 2005 Jun;128(7):2119-23. doi: 10.1053/j.gastro.2004.12.035. PMID 15940642
- [Background] Sasajima K, Kudo SE, Inoue H, Takeuchi T, Kashida H, Hidaka E, Kawachi H, Sakashita M, Tanaka J, Shiokawa A. Real-time in vivo virtual histology of colorectal lesions when using the endocytoscopy system. Gastrointest Endosc. 2006 Jun;63(7):1010-7. doi: 10.1016/j.gie.2006.01.021. PMID 16733118
- [Background] Eberl T, Jechart G, Probst A, Golczyk M, Bittinger M, Scheubel R, Arnholdt H, Knuechel R, Messmann H. Can an endocytoscope system (ECS) predict histology in neoplastic lesions? Endoscopy. 2007 Jun;39(6):497-501. doi: 10.1055/s-2007-966446. PMID 17554643
- [Background] Cipolletta L, Bianco MA, Rotondano G, Piscopo R, Meucci C, Prisco A, Cipolletta F, de Gregorio A, Salvati A. Endocytoscopy can identify dysplasia in aberrant crypt foci of the colorectum: a prospective in vivo study. Endoscopy. 2009 Feb;41(2):129-32. doi: 10.1055/s-0028-1103452. Epub 2009 Feb 12. PMID 19214891
- [Background] Rotondano G, Bianco MA, Salerno R, Meucci C, Prisco A, Garofano ML, Sansone S, Cipolletta L. Endocytoscopic classification of preneoplastic lesions in the colorectum. Int J Colorectal Dis. 2010 Sep;25(9):1111-6. doi: 10.1007/s00384-010-0969-7. Epub 2010 Jun 8. PMID 20532533
- [Background] Neumann H, Fuchs FS, Vieth M, Atreya R, Siebler J, Kiesslich R, Neurath MF. Review article: in vivo imaging by endocytoscopy. Aliment Pharmacol Ther. 2011 Jun;33(11):1183-93. doi: 10.1111/j.1365-2036.2011.04647.x. Epub 2011 Apr 4. PMID 21457290